CLINICAL TRIAL: NCT04545645
Title: The Effect of Auditory and Motor Cognitive Distractions on the Neural Provocation Test in Subjects With Neck Pain: A Randomized Controlled Trial
Brief Title: The Effect of Auditory and Motor Cognitive Distractions on the Neural Provocation Test in Subjects With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: uammadrid30
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Neural Stress Provoked by the Median Nerve (Active Comparator)
  Interventions: Behavioral: median nerve mobilization
- Neural stress provocation with cognitive auditory distraction (Experimental)
  Interventions: Behavioral: Neural stress provocation with cognitive auditory distraction
- Providing neural stress with a motor distraction (Experimental)
  Interventions: Behavioral: Providing neural stress with a motor distraction
- Neural stress provocation with both distractions (Experimental)
  Interventions: Behavioral: Neural stress provocation with auditory and motor cognitive distraction.

INTERVENTIONS:
Behavioral: median nerve mobilization — The patient is placed in a supine position and his cervical spine with 25º of lateral flexion on the opposite side of the member in which we perform the test. First a passive scapular depression is performed, 90º of shoulder abduction combining external shoulder rotation. Next, a supination of the forearm is performed with wrist extension and finger extension. Finally, the elbow is extended to the limit of resistance or when the investigator observes the elevation of the shoulder girdle.
  Arms: Neural Stress Provoked by the Median Nerve
Behavioral: Neural stress provocation with cognitive auditory distraction — Neural provocation of the median nerve is performed but an auditory distraction is added with a metronome with a constant time of 50 beats per minute.
  Arms: Neural stress provocation with cognitive auditory distraction
Behavioral: Providing neural stress with a motor distraction — The neural provocation of the median nerve is performed and we add a motor distraction that consists of the patient intermittently squeezing a ball with the opposite hand.
  Arms: Providing neural stress with a motor distraction
Behavioral: Neural stress provocation with auditory and motor cognitive distraction. — The neural provocation of the median nerve is performed, we add auditory distraction with the metronome with a constant time of 50 BPM and a motor distraction consisting of squeezing a ball to the rhythm that sounds the metronome.
  Arms: Neural stress provocation with both distractions

SUMMARY:
The main objective of this research is to evaluate the influence of different distraction stimuli on neural mechano-sensitivity tests.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 65 years
* Medical diagnosis of non specific chronic neck pain with more than 6 months of evolution of neck pain

Exclusion Criteria:

* Patients with rheumatic diseases, cervical hernia, cervical whiplash syndrome, neck surgeries o a history of arthrodesis
* Systemic diseases
* Vision, hearing or vestibular problems
* Severe trauma or a traffic accident that had an impact on the cervical area.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Mechanosensitivity based on range of motion | Change in pressure pain threshold immediately at the end of the intervention
  The inclinometer, an instrument characterized by the constant use of gravity as a reference point to evaluate mobility, is used to evaluate the range of nerve movement.
Pain intensity | Change in pain intensity immediately at the end of the intervention
  It is the subjective feeling of self-reported pain ranging from 0-100 points.

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain